CLINICAL TRIAL: NCT06399510
Title: Electrolyte Balance Effects of Sterofundin Versus Normal Saline in Diabetic Ketoacidosis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Sains Malaysia (Other)
Responsible Party: Principal Investigator, Mohd Zulfakar Mazlan, MBBS, Associate Professor, Universiti Sains Malaysia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: USM/JEPeM/KK/23100751
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-03 (Actual); Status verified 2024-04

CONDITIONS: Treatment Diabetic Ketoacidosis, Electrolyte Balance Effects

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal Saline (Active Comparator): If patients were randomized to the control arm, the fluid regime for the first 24 hours in ICU will be normal saline.
  Interventions: Other: Sterofundin fluid therapy
- Sterofundin (Experimental): If patients were randomized to the interventional arm, the main fluid therapy during the first 24 hours of ICU stay will be Sterofundin.
  Interventions: Other: Sterofundin fluid therapy

INTERVENTIONS:
Other: Sterofundin fluid therapy — Sterofundin is known as balanced solution which has similar electrolytes content as per human plasma.

SUMMARY:
The goal of this prospective single centered randomized control trial is to compare the electrolyte balance effects between Sterofundin and Normal Saline in Diabetic Ketoacidosis patients. The main questions it aims to answer are:

i. Is there any difference in duration of bicarbonate (HCO3-) to reach equal or more than 15mmol/L from the initial blood taking in between Sterofundin and NS fluid use in DKA patients? ii. Is there any difference in the level of post-infusion serum sodium (Na+) between Sterofundin and NS fluid use in DKA patients? iii. Is there any difference in the level of post-infusion serum potassium (K+) between Sterofundin and NS fluid use in DKA patients?

Patients will be randomized in a 1:1 ratio to receive IV Sterofundin (intervention) or IV Normal Saline (standard care). The patient will have the respective fluid regime as the main fluid therapy during the first 24 hours of ICU stay. If patients were randomized to the control arm, the fluid regime for the first 24 hours in ICU will be normal saline. If patients were randomized to the interventional arm, the main fluid therapy during the first 24 hours of ICU stay will be Sterofundin.

ELIGIBILITY:
Inclusion Criteria:

* DKA.
* Aged ≥ 18 years old.
* Patients admitted to ICU < 12 hours after initial fluid resuscitation from emergency department/ ward.

Exclusion Criteria:

* End stage renal failure
* Heart failure
* Started treatment of sodium bicarbonate infusion prior to ICU admission
* Known allergy to Sterofundin

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
The duration taken for serum HCO3 ≥ 15 within 24 hours ICU admission. | 24 Hours
Mean difference of serum sodium level between Sterofundin and normal saline fluid use in diabetic ketoacidosis patients | 24 Hours
Mean difference of serum potassium level between Sterofundin and normal saline fluid use in diabetic ketoacidosis patients. | 24 Hours

SECONDARY OUTCOMES:
The Need of Renal Replacement Therapy | 30 days
Mechanical ventilation day | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universiti Sains Malaysia, Kubang Kerian, Kelantan, Malaysia

IPD SHARING:
Plan to Share IPD: No